CLINICAL TRIAL: NCT05669001
Title: A 12-Month, Randomized, Open-Label, Phase IIA Study Evaluating the Safety and Efficacy of Siplizumab in Combination With Belatacept and MPA Compared to Standard of Care Immunosuppression in de Novo Renal Transplant Recipients (ASCEND)
Brief Title: A Study of TCD601 in de Novo Renal Transplant Recipients
Acronym: ASCEND
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCD601B203
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — siplizumab; Abatacept; Antilymphocyte Serum; Tacrolimus; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TCD601 (siplizumab) (Experimental): TCD601 administered in combination with belatacept, mycophenolic Acid (MPA), and corticosteroids
  Interventions: Biological: TCD601; Biological: belatacept; Drug: MPA; Drug: Corticosteroids
- ATG (Active Comparator): Antithymocyte globulin (ATG), tacrolimus (TAC), mycophenolic acid (MPA), and corticosteroids
  Interventions: Drug: ATG; Drug: TAC; Drug: MPA; Drug: Corticosteroids

INTERVENTIONS:
Biological: TCD601 — Investigational Product
  Other Names: siplizumab
  Arms: TCD601 (siplizumab)
Biological: belatacept — Study Product
  Arms: TCD601 (siplizumab)
Drug: ATG — Comparator
  Other Names: antithymocyte globulin
  Arms: ATG
Drug: TAC — Comparator
  Other Names: tacrolimus
  Arms: ATG
Drug: MPA — Immunosuppression Therapy
  Other Names: mycophenolic acid
Drug: Corticosteroids — Immunosuppression Therapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TCD601 in combination with Belatacept when compared to standard of care immunosuppression therapy in de novo renal transplant patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of TCD601 (siplizumab), an anti-CD2 monoclonal antibody, in combination with a CNI-free regimen of belatacept, MPA, and corticosteroids compared to a standard of care CNI-based regimen of tacrolimus, ATG, MPA and corticosteroids in de novo renal transplant patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand the study requirements and provide written informed consent before and study assessment is performed
* Male or female patients ≥ 18 to 70 years of age
* Recipients of a de novo renal allograft from a heart-beating deceased, living ABO compatable, non-HLA identical living related donor

Key Exclusion Criteria:

* Subjects who have received a kidney allograft previously
* Recipient of a kidney from an HLA identical living related donor
* Recipient of a kidney from a donor after cardiac death

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs) and serious adverse events (SAEs) in Arm 1 compared to Arm 2 | 12 months
  The number of adverse events and serious adverse events

SECONDARY OUTCOMES:
Renal function in Arm 1 compared to Arm 2 | 12 months
  renal function using estimated glomerular filtration rate (eGFR)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Juhlin, Study Director — ITB-Med LLC
Locations (17):
- United States (17):
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia Health, Charlottesville, Virginia
  - Inova Fairfax Hospital Medical Campus, Falls Church, Virginia